CLINICAL TRIAL: NCT03685929
Title: Histopathological Comparison Between Superficial Pressure Ulcers and Incontinence-associated Dermatitis
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/0946
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Pressure Ulcer; Incontinence-associated Dermatitis; Irritant Contact Dermatitis; Diaper Rash
Keywords: Pressure ulcer; Incontinence-associated dermatitis; Histopathology; Ischemia; Irritation; Prevention; Tissue; Skin
MeSH Terms: conditions — Pressure Ulcer; Dermatitis, Irritant; Diaper Rash; Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Punch skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pressure ulcers: Patients with pressure ulcers category II/III at sacrum or trochanter
  Interventions: Procedure: Punch skin biopsy
- Incontinence-associated dermatitis: Patients with incontinence-associated dermatitis category IIA at sacrum (or trochanter)
  Interventions: Procedure: Punch skin biopsy
- Combined lesion: Patients with pressure ulcer category II/III and incontinence-associated dermatitis category IIA at sacrum or trochanter
  Interventions: Procedure: Punch skin biopsy

INTERVENTIONS:
Procedure: Punch skin biopsy — Two punch biopsies will be performed in each patient, one at the border of the skin lesion, and one at the adjacent healthy skin. A disposable biopsy punch of 4 mm will be used. A biopsy punch is a small circular blade (like an apple corer) which is rotated into the skin to obtain a cylindrical specimen. Local anaesthesia will be applied and the circular wound will be closed by a single suture. Sutures will be removed after one week.

SUMMARY:
This study aims to identify differences and similarities between superficial pressure ulcers (category II and III) and incontinence-associated dermatitis (category IIA) at tissue level.

Skin biopsies will be obtained from 30 patients with pressure ulcers (n = 10), incontinence-associated dermatitis (n = 10), and combined lesions (n = 10).

The results from the histopathologic examination will be compared with the clinical diagnosis by wound care experts, which will be based on photographs and relevant patients' characteristics.

DETAILED DESCRIPTION:
Despite current preventive strategies, prevalence of pressure ulcers and incontinence-associated dermatitis (IAD) is still estimated at 5.9-6.9% in hospitalised patients, and 5.0-5.9 in home care patients. Both skin conditions may occur in the same body region but are considered as separate entities, based on differences in etiology.

At tissue level, it is assumed that pressure ulcers are characterised by ischemia and tissue deformation. In contrast, IAD is assumed to be characterised by an irritative pattern. These assumptions are reflected in current preventive strategies. However, a small scale study, performed by Houwing et al. (2007), described the additional presence of an ischemic pattern in patients with IAD. More insights into the histopathologic pattern of pressure ulcers and IAD is needed to optimise current preventive strategies.

Tha aim of this study is to compare superficial pressure ulcers (category II and III) and IAD (category IIA) at tissue level.

A prospective interventional study will be performed during which skin biopsies (punch biopsies) will be collected from 30 incontinent patients. In each patient patient, two punch skin biopsies will be performed, one at the border of the skin lesion and one at the adjacent healthy skin. Sections from the biopsies will be stained with hematoxiline and eosine and examined by two independently working, blinded skin pathologists. In addition, photographs from the skin lesions will be analysed by 10 national and international wound care experts to promote correct diagnosis. Finally, findings from the histopathologic examination will be compared with the clinical diagnoses based on photographs.

ELIGIBILITY:
Inclusion Criteria:

* Incontinent for urine, stool, or both
* Superficial pressure ulcer (category II or III) and/or incontinence-associated dermatitis (category IIA)
* Expected length of stay of 7 days following punch skin biopsy

Exclusion Criteria:

* Skin infection at biopsy site
* Medical contraindication to obtain a biopsy
* End of life care
* Not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted on following wards of a university hospital
  * Pneumology
  * Gastroenterology
  * Endocrinology
  * Nephrology
  * Neurology
  * Geriatrics
  * Gastrointestinal surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of pressure ulcers and incontinence-associated dermatitis | 1 day
  Presence of pressure ulcers and/or incontinence-associated dermatitis based on photographs and patient characteristics
Histopathologic pattern | 1 day
  Characteristics of epidermis, dermis, and subcutis based on histopathologic examination

SECONDARY OUTCOMES:
Rate of agreement between visual and histopathologic diagnosis | 1 day
  Agreement between diagnosis of wound care experts (based on photographs), and diagnosis by skin pathologists (based on histopathologic examination)

CONTACTS AND LOCATIONS:
Overall Officials: Sofie De Schepper, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beeckman D, Van Damme N, Schoonhoven L, Van Lancker A, Kottner J, Beele H, Gray M, Woodward S, Fader M, Van den Bussche K, Van Hecke A, De Meyer D, Verhaeghe S. Interventions for preventing and treating incontinence-associated dermatitis in adults. Cochrane Database Syst Rev. 2016 Nov 10;11(11):CD011627. doi: 10.1002/14651858.CD011627.pub2. PMID 27841440
- See also: Website of the research group — http://www.UCVVGent.be